CLINICAL TRIAL: NCT06959316
Title: Pregnancy Data Repository to Assess Management of Type 1 Diabetes With Diabetes Technology
Brief Title: T1D Pregnancy & Me
Acronym: PRAM-T1D
Status: Recruiting | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Other Study IDs: PRAM-T1D
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 1; Pregnancy in Diabetics; Pregnancy, High-Risk; Insulin Dependent Diabetes
Keywords: Type 1 diabetes; Pregnant; Pregnancy; Insulin pump; Continuous glucose monitor; Remote study; Online study; T1D; CGM; Insulin injection; Hybrid closed loop; HCL
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pregnancy in Diabetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCL Use: Pregnant individuals with type 1 diabetes (T1D) using HCL systems for glycemic management in pregnancy
  Interventions: Device: Hybrid closed loop insulin delivery system
- HCL Non-Use: Pregnant individuals with type 1 diabetes (T1D) not using HCL systems for glycemic management in pregnancy

INTERVENTIONS:
Device: Hybrid closed loop insulin delivery system — Hybrid closed loop insulin delivery system is a system that uses a continuous glucose monitor (CGM) to send blood glucose values to an insulin pump that automatically provides insulin based on the blood glucose value and anticipated future level.
  Groups: HCL Use

SUMMARY:
T1D Pregnancy & Me will partner with pregnant participants living with type 1 diabetes (T1D) in the United States to collect real-world data on management of T1D in pregnancy. This is a remote study where participants can complete online surveys and share device data (continuous glucose monitor (CGM) data and insulin data). Through the collection of CGM, insulin, and pregnancy outcome data, the study will provide important information to understand how diabetes is being managed during pregnancy. These data will provide much needed evidence to guide modern management of diabetes during pregnancy with a goal of improving care and outcomes.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) management during pregnancy is a critical area as pregnancy complicated by T1D is still associated with a markedly elevated risk of maternal and fetal complications. Because the risk of these complications is tightly linked to glucose levels, guidelines recommend lower glycemic targets than in non-pregnant individuals to optimize pregnancy outcomes. Hybrid closed loop (HCL) insulin delivery systems may aid in glycemic management during pregnancy, but options for use of HCL during pregnancy are limited and present challenges as systems are not approved for use in pregnancy and do not target pregnancy glycemic goals. Thus, pregnant individuals with T1D and their clinicians must consider off-label use of HCL systems with suboptimal glycemic targets. To get closer to pregnancy glycemic targets, individuals may adjust the way they use the system, but there is insufficient evidence to understand the impact of HCL systems available in the US on pregnancy glycemic metrics and pregnancy outcomes.

To address these gaps in evidence, we propose an observational study that will enable systematic assessment of HCL system use in pregnancies complicated by T1D. The focus of this study is to assess glycemic outcomes measured by continuous glucose monitors and clinical pregnancy outcomes associated with use of HCL versus other insulin delivery methods. Data collected from this study will provide important information about how individuals in the United States are managing their diabetes during pregnancy and will help us to identify factors that could minimize the risk of diabetes-associated pregnancy complications and reduce the burden that comes with managing T1D in pregnancy.

Pregnant individuals throughout the United States will be enrolled in this remote observational study. Participants will be asked to share details about their diabetes and pregnancy. Participants will also be asked to share diabetes device data from their continuous glucose monitor (CGM). Participants who use an insulin pump or connected insulin pen may also be asked to share these data.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Clinical diagnosis of presumed T1D for at least 6 months duration
3. Less than 15 weeks gestation at time of enrollment based on due date from provider
4. Planned CGM use on a regular basis (e.g., ≥10 out of 14 days) and willing to continue using CGM regularly with no plans to discontinue CGM use during the study
5. Following intensive insulin therapy regimen defined as basal-bolus delivery via an insulin pump (including a closed loop system) or multiple daily injections (MDI)
6. Have access to technology that may be required to complete study questionnaires and share diabetes device data.
7. Resident of the United States and plans to reside in the U.S. for the duration of the study
8. Comprehends written and spoken English or Spanish
9. Willing and able to provide informed consent, complete surveys and provide the device data that are part of the protocol

Exclusion Criteria:

1. Multiple pregnancy
2. Current renal dialysis or plan to begin renal dialysis during the study
3. History of liver cirrhosis
4. Active cancer treatment with systemic chemotherapy
5. Current participation in other studies involving an investigational insulin delivery device or planning to participate in an investigational insulin delivery device study during pregnancy
6. Prior participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant adults with type 1 diabetes from across the United States who use a continuous glucose monitor.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
CGM Outcome (BG 63-140 mg/dl) | Up to 37 weeks gestation
  Percentage of time spent with glucose 63-140 mg/dl

SECONDARY OUTCOMES:
CGM Outcome (BG<63 mg/dl) | Up to 37 weeks gestation
  Percentage time spent with glucose <63 mg/dl
CGM Outcome (BG<54 mg/dl) | Up to 37 weeks gestation
  Percentage time spent with glucose <54 mg/dl
CGM Outcome (BG>140 mg/dl) | Up to 37 weeks gestation
  Percentage time spent with glucose >140 mg/dl

OTHER OUTCOMES:
Hypertensive disorder of pregnancy | Up to 37 weeks gestation
  Gestational hypertension or preeclampsia
LGA Status (defined as birthweight percentile > 90th) | At birth
  Large gestational age birthweight
Preterm delivery | Delivery after 20 weeks and before 37 weeks gestation
  Preterm delivery
Neonatal Morbidity | At birth
  Hypoglycemia, hyperbilirubinemia, respiratory distress, or birth trauma

CONTACTS AND LOCATIONS:
Overall Officials: Robin Gal, MSPH, Principal Investigator — Jaeb Center for Health Research; Camille Powe, MD, Study Chair — Massachusetts General Hospital
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barbara Davis Center for Diabetes & University of Colorado Health, Aurora, Colorado
  - Jaeb Center for Health Research, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - Mass General Brigham, Boston, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided